CLINICAL TRIAL: NCT04129138
Title: A Survey of High Risk Patient and Caregiver Attitudes and Beliefs Regarding the Prescription of Intranasal Naloxone Spray for Opioid Overdose
Brief Title: Patient and Caregiver Attitudes and Beliefs Regarding Prescription of Intranasal Naloxone Spray for Opioid Overdose
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2019-0330; NCI-2019-06740 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0330 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Caregiver; Patient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (survey): Participants complete a survey over 30 minutes.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete survey

SUMMARY:
This trial studies the attitudes and beliefs of high risk patients and caregivers regarding the prescription of intranasal naloxone spray for opioid overdose. Knowledge regarding high risk patients' and caregivers' beliefs and attitudes regarding co-prescription of naloxone spray with opioids may help to identify barriers to prescribing and helping tailor the education to better meet the needs of patients and caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the proportion of high risk patients who perceive receiving a prescription of intranasal naloxone to be beneficial for them.

SECONDARY OBJECTIVES:

I. To determine the proportion of caregivers who perceive receiving a prescription of intranasal naloxone to be beneficial for the patient.

II. To determine the association between high risk patients' and their caregivers' characteristics (this includes cut-annoyed-guilty-eye [CAGE], screener and opioid assessment for patients with pain [SOAPP], age, gender, ethnicity, education, employment status, presence of caregiver, cancer type, cancer stage, reason for Narcan prescription, health insurance, and setting of Narcan prescription) and their perception that a prescription for intranasal naloxone is beneficial for patients.

EXPLORATORY OBJECTIVE:

I. To conduct an exploratory analysis of high risk patients' and caregivers' attitudes and beliefs regarding prescription of intranasal naloxone spray.

OUTLINE:

Participants complete a survey over 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been prescribed intranasal naloxone in the past 1 year
* Patients and caregivers must be able to understand, read, write, and speak English
* Patients must have no clinical evidence of cognitive impairment, as determined by the palliative care provider (Memorial Delirium Assessment Scale score of >= 7)
* Patients must sign an informed consent
* Caregivers may sign an informed consent if available during the visit
* Caregivers may verbally consent over the phone if not present during the visit
* Caregiver must be a friend, significant other or family member
* Caregivers must have no evidence of cognitive impairment, as determined based on orientation questions pertaining to the date, day of the week, time, and place

Exclusion Criteria:

* PATIENT: Emotional or psychosocial distress as identified by the patient's palliative care
* PATIENT: Participants with Edmonton Symptom Assessment System (ESAS) anxiety score of > 6

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients prescribed naloxone in the last year and their caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2020-07-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To determine the proportion of high risk patients who perceive receiving a prescription of intranasal naloxone to be beneficial for them | Up to 1 year

SECONDARY OUTCOMES:
To determine the proportion of caregivers who perceive receiving a prescription of intranasal naloxone to be beneficial for the patient. | Up to 1 year
To determine the association between high risk patients' and their caregivers' characteristics | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jaya S Amaram-Davila, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org